CLINICAL TRIAL: NCT06940180
Title: Perioperative Chemoimmunotherapy With Toripalimab for Sinonasal Cancer
Brief Title: Toripalimab With Chemotherapy for Sinus Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn J. Hanna (Other)
Collaborators: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Glenn J. Hanna, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-121
Record Dates: First submitted 2025-04-09; First posted 2025-04-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Sinonasal Cancer; Paranasal Sinus Neoplasms; Squamous Cell Carcinoma; Sinonasal Undifferentiated Carcinoma; Locally Advanced Head and Neck Cancer
Keywords: Paranasal Sinus Neoplasm; Squamous Cell Carcinoma; Sinonasal Undifferentiated Carcinoma; Locally Advanced Head and Neck Cancer; Advanced Sinonasal Cancer; Advanced Paranasal Sinus Cancer; Sinonasal Cancer
MeSH Terms: conditions — Paranasal Sinus Neoplasms; Carcinoma, Squamous Cell; Sinonasal undifferentiated carcinoma; Head and Neck Neoplasms | interventions — toripalimab; Carboplatin; Docetaxel; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Toripalimab and Docetaxel Plus Carboplatin (TCD) (Experimental): * Baseline visit with imaging
  * Cycles 1 and 2 (21 day cycles)
    * Day 1: Predetermined dose of Toripalimab 1x daily
    * Day 1: Chemotherapy: predetermined dose of Docetaxel 1x daily and Carboplatin 1x daily
  * Tumor assessment by imaging
  * Surgical resection of tumor
  Interventions: Drug: Toripalimab; Drug: Carboplatin; Drug: Docetaxel
- Arm 2: Post Operative Radiation Therapy + Toripalimab (Experimental): After pathology assessment, participants with a pathological treatment response of 2 will be assigned radiation therapy per standard practice guidelines and predetermined dose of Toripalimab 1x every 3 weeks for up to 8 cycles (21 day cycles).
  -Follow up: every 3 months for 1 year. Imaging at 3 months
  Interventions: Drug: Toripalimab; Radiation: Radiation Therapy
- Arm 3: Post Operative Radiation Therapy With or Without Chemotherapy (Experimental): After pathology assessment, participants with a pathological treatment response of 2 or less will be assigned standard radiation therapy with or without standard of care Cisplatin-based chemotherapy as recommended per treatment team and standard practice guidelines.
  -Follow up: every 3 months for 1 year. Imaging at 3 months
  Interventions: Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Toripalimab — An anti-PD-1 monoclonal antibody, single-use vial, via intravenous (into the vein) infusion per protocol.
  Other Names: TAB-001; JS001; CHS-007; Loqtorzi; Toripalimab-tpzi
  Arms: Arm 1: Toripalimab and Docetaxel Plus Carboplatin (TCD); Arm 2: Post Operative Radiation Therapy + Toripalimab
Drug: Carboplatin — An antineoplastic agent, multi-dose vials, via intravenous (into the vein) infusion per standard of care.
  Arms: Arm 1: Toripalimab and Docetaxel Plus Carboplatin (TCD)
Drug: Docetaxel — A taxoid antineoplastic agent, single-dose vials, via intravenous (into the vein) infusion per standard of care.
  Other Names: Docefrez; Taxotere; C43H53NO14∙3H2O
  Arms: Arm 1: Toripalimab and Docetaxel Plus Carboplatin (TCD)
Radiation: Radiation Therapy — per standard of care
  Arms: Arm 2: Post Operative Radiation Therapy + Toripalimab; Arm 3: Post Operative Radiation Therapy With or Without Chemotherapy
Drug: Cisplatin — An antineoplastic agent, single-dose vials, via intravenous (into the vein) infusion per standard of care.
  Other Names: Cl2H6N2Pt; Platinol; Platinol-AQ
  Arms: Arm 3: Post Operative Radiation Therapy With or Without Chemotherapy

SUMMARY:
The aim of this research study is to evaluate the effectiveness and safety of a combination of immunotherapy, using a drug called toripalimab, with chemotherapy drugs, Carboplatin and Docetaxel, as a possible treatment before surgery for sinonasal cancers.

The names of the study drugs used in this research study are:

* Toripalimab (a type of monoclonal antibody)
* Carboplatin (a type of antineoplastic agent)
* Docetaxel (a type of antineoplastic agent)
* Cisplatin (a type of antineoplastic agent)

DETAILED DESCRIPTION:
This single-arm, open-label, single-center phase II study is to evaluate the effectiveness and safety of a combination of immunotherapy, using a drug called toripalimab with chemotherapy drugs, Carboplatin and Docetaxel, as a possible treatment before surgery for sinonasal cancers.

Toripalimab binds to the PD-1 receptors on T-cells (immune cells) and prevents them from interacting with PD-L1 and PD-L2 on tumor cells. This stimulates the immune system to fight tumor cells.

The U.S. Food and Drug Administration (FDA) has not approved Toripalimab for sinonasal cancers, but it has been approved for another type of head and neck cancer called nasopharyngeal carcinoma (NPC), in the advanced incurable setting when surgery is no longer possible, or when cancer has spread to parts of the body outside the head and neck region.

Carboplatin and Docetaxel have been approved by the FDA in the advanced incurable setting for other types of head and neck cancer.

The research study procedures include screening for eligibility, in-clinic visits, questionnaires, blood tests, urine tests, X-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission (PET) scans, and photographic images of tumors.

It is expected that about 20 people will take part in this research study.

Coherus Biosciences, a pharmaceutical company, is funding this research study by providing the study drug and funding for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed locoregionally advanced nasal cavity or paranasal sinus cancer including the following histologic subtypes: squamous cell carcinoma (SCC) of any morphologic variation: verrucous, papillary, basaloid, spindle cell, and adenosquamous; or sinonasal undifferentiated carcinoma (SNUC).
* Participants with SCC should have resectable disease at baseline per the discretion of the treating surgical oncologist(s). *Participants with SNUC can have operable or borderline resectable (definition: resection would been morbid requiring extensive surgery and would have chances of incomplete gross total resection) disease as judged by the treating surgical oncologist(s).
* Participants must have clinical stage disease as defined below using the 8th (2017) edition of the tumor, node, metastasis (TNM) staging system by the American Joint Committee on Cancer (AJCC) and the Union for International Cancer Control (UICC):

  * T2, N1-3 III
  * T3, any N III, IVA, IVB
  * T4, any N IVA, IVB
* Participants must be willing to provide blood and tissue pre-treatment and at the time of surgery for pathologic and correlative analyses.
* Age 18 years or older at the time of informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥1000/mcL
  * Platelets ≥100
  * Total bilirubin ≤institutional upper limit of normal (ULN)
  * AST(SGOT) / ALT (SGPT) ≤3x ULN
  * Creatinine ≤institutional ULN or GFR of ≥50 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Contraception use should be maintained until at least 6 months after the last dose of chemotherapy for females and 3 months for males. In addition, contraception use should continue until 4 months after last dose of toripalimab for both males and females.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with nasal cavity or paranasal sinus malignancies demonstrating histologies other than SCC or SNUC in the opinion of the reviewing pathologist. Excluded subtypes include: angiosarcomas, rhabdomyosarcomas, lymphomas, olfactory neuroblastomas (esthesioneuroblastomas), melanomas, and meningiomas among others. SNEC or sinonasal neuroendocrine carcinoma is not permitted.
* Participants with unresectable or inoperable disease as judged by the treating surgical oncologist(s).
* Participants with known distant metastatic disease (M1 or IVC).
* Has received prior therapy with an anti-PD-1/L1 agent or any other agent directed to another stimulatory or co-inhibitory T-cell receptor.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Non-live vaccines are permitted.
* Carries a diagnosis of immunodeficiency or is receiving chronic systemic corticosteroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Exceptions may be permitted at the discretion of the overall Sponsor-Investigator.
* Has an active autoimmune disease that has required systemic treatment in past 6 months (with use of a disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is permitted.
* Has a history of (non-infectious) pneumonitis or interstitial lung disease that required steroids or has current pneumonitis or interstitial lung disease.
* Has a known history of human immunodeficiency virus (HIV) infection that is uncontrolled. No HIV testing is required unless mandated by local health authority. Patients with well controlled HIV may be eligible if their CD4 T cell count is favorable and their HIV viral load is undetectable.
* Has a known history of active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a history of allogeneic tissue or solid organ transplant.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Treatment Response Rate (pTRR) | Tumor assessments or scans will be obtained at baseline and 3-months following the end of treatment. Treatment duration is not fixed and this observation time is variable, criteria for discontinuation is outlined in protocol section 5.10.
  pTRR is defined as the proportion of participants that experience a complete pathologic response or partial pathologic response during treatment, as defined in the RECIST criteria.

SECONDARY OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | Adverse events are collected every study visit through study completion, an average of 1 year. Treatment duration is not fixed and this observation time is variable, criteria for discontinuation is outlined in protocol section 5.10.
  Safety and tolerability assessed by CTCAE v5.0 and summarized descriptively.
Median Disease-free Survival (DFS) | Tumor assessments or scans will be obtained at baseline and 3-months following the end of treatment. Treatment duration is not fixed and this observation time is variable, criteria for discontinuation is outlined in protocol section 5.10.
  Disease-free survival (PFS) is defined as the time from the date of study registration to first invasive local, regional, distant recurrence, or death due to any cause. Participants alive without disease are censored at date of last disease evaluation.
Median Overall Survival (OS) | Participants will be followed for 1-year (12 months) after completion or removal from protocol therapy or until death, whichever occurs first. Treatment duration is not fixed and this observation time is variable, criteria for discontinuation is outlined
  OS is Overall survival based on the Kaplan-Meier method is defined as the time from randomization to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Organ Preservation Rate | Up to 42 days.
  Defined as the percentage of patients with an intact orbit, palate, and skull base immediately post-op from definitive oncologic resection among the study cohort.
Overall Response Rate (ORR) | Up to 42 days.
  ORR is the proportion of participants that experience complete response (CR) or partial response (PR) recorded from the start of the TCD treatment to the first imaging just prior to surgery.
Correlation between tumor PD-L1 combined positive score (CPS) with pTR | Tumor assessments or scans will be obtained at baseline and 3-months following the end of treatment. Treatment duration is not fixed and this observation time is variable, criteria for discontinuation is outlined in protocol section 5.10
  PD-L1 CPS values range from 0-100. Higher scores are considered positive.
Correlation between tumor PD-L1 combined positive score (CPS) with survival outcomes | Participants will be followed for 1-year (12 months) after completion or removal from protocol therapy or until death, whichever occurs first. Treatment duration is not fixed and this observation time is variable per protocol.
  PD-L1 CPS values range from 0-100. Higher scores are considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu